CLINICAL TRIAL: NCT06420674
Title: Online Prevention of Emotional Disorders in Women Undergoing Fertility Treatments (RE-FER Moodle)
Brief Title: Online Prevention of Emotional Disorders in Women Undergoing Fertility Treatments
Acronym: RE-FER moodle
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jorge Javier Osma López (Other)
Collaborators: Hospital General Universitario de Castellón (Other); Hospital Universitario La Plana de Castellón (Unknown)
Responsible Party: Sponsor-Investigator, Jorge Javier Osma López, Associate Professor, Instituto de Investigación Sanitaria Aragón
Organization: Instituto de Investigación Sanitaria Aragón (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IPES/RE-FER/moodle
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Infertility; Emotional Disorder; Anxiety Depression
Keywords: Unified Protocol; Prevention; Anxiety; Depression; Reproduction
MeSH Terms: conditions — Infertility; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: This study will be offered to all women undergoing artificial inseminations in two public hospitals.
Masking Description: Masking is not applicable in this study as it includes only one condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RE-FER web (Experimental): The study will be offered to all women receiving artificial inseminations in two Spanish public hospitals (Hospital Universitario General de Castellón and Hospital Universitario La Plana).
  Interventions: Behavioral: Unified Protocol for Transdiagnostic Treatment of Emotional Disorders

INTERVENTIONS:
Behavioral: Unified Protocol for Transdiagnostic Treatment of Emotional Disorders — The Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders is a psychological intervention that focuses on a wide range of emotional disorders (i.e., anxiety, depression and related disorders). It allows care for comorbid disorders, subclinical or unspecified symptoms reducing associated costs and improving response to treatment.
  In our study, the Unified Protocol preventive program will be applied throughout 10 online modules. Women will have access to a web-page (moodle version) that includes audiovisual materials (e.g., written manual, videos, editable registers) and psychological assessments.

SUMMARY:
The main aim of this pilot study is to study the clinical utility and acceptability of a transdiagnostic psychological intervention, the Unified Protocol, delivered in online format to prevent the onset of emotional disorders in a sample of women undergoing fertility treatments (artificial insemination). The main questions it aims to answer are:

1. Can the Unified Protocol help to prevent the onset of emotional disorders during fertility treatments? The investigators expect to find a maintenance or improvement in anxiety and depressive symptoms as well as on quality of life and fertility-related stress.
2. Would the Unified Protocol delivered in online format be well accepted by women undergoing fertility treatments? The investigators expect to find high satisfaction rates both with the Unified Protocol contents and the online format.

DETAILED DESCRIPTION:
Women who can not achieve a spontaneous pregnancy (i.e., couples who had fertility problems, single women or same-sex couples) frequently ask for fertility treatments. These treatments can provide the opportunity to get the desired pregnancy. However, they are also experienced as a highly stressful situation which has a direct impact on women's lives. It has been reported that fertility treatments are associated with high levels of stress, worse quality of life, high interference with women's life and the development of emotional disorders such as anxiety and depression. Between 25 and 65% of women undergoing fertility treatments suffer from anxiety and depressive symptoms, frequently with high comorbidity rates between these two psychological conditions. Also worrisome, these emotional disorders are one of the most notable reasons to discontinue fertility treatments.

In this scenario, different national and international organizations have postulated the need to implement psychological assessments and interventions in women undergoing fertility treatments. However, some personal (i.e., lack of time) and logistical barriers (i.e., lack of psychologist in Human Reproduction Units and high distances to the hospital), impede that these psychological programs are finally implemented in Human Reproduction Units.

New Information and Communication Technologies have been widely developed to provide psychological care in populations suffering emotional disorders, even in women undergoing fertility treatments. However, these technology-based solutions have not been yet implemented in the Spanish national healthcare system.

According to this information, the purpose of this study is to explore the clinical utility and acceptability of a web-based transdiagnostic psychological intervention, the Unified Protocol, to prevent the onset of anxiety and depressive symptoms in women undergoing artificial inseminations.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age.
* Have a good understanding of Spanish.
* Have started fertility treatment (at least one artificial insemination received).
* Signed the informed consent.

Exclusion Criteria:

* Not having Internet access to access the web-page.
* Having a diagnosis of severe mental disorder.
* Active suicidal ideation at the time of evaluation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Overall Depression Severity and Impairment Scale (ODSIS) | Pre-intervention; Post-intervention, 11 weeks from pre-assessment; 1 month follow-up after post-assessment; 3 months follow-up after post-assessment; 6 months follow-up after post-assessment.
  This questionnaire consist of 5 items that evaluate the frequency and the intensity of depressive symptoms and their interference in life (e.g., work, school and social life). It is responded on a 5-point Likert scale (0=No depression - 4=The worst depression possible). The total score range from 0 to 20 points. Higher scores are indicative of greater severity and functional impairment as a result of depressive symptoms. In the Spanish population the clinical cut-off has been stablished in 10 points.
Overall Anxiety Severity and Impairment Scale (OASIS) | Pre-intervention; Post-intervention, 11 weeks from pre-assessment; 1 month follow-up after post-assessment; 3 months follow-up after post-assessment; 6 months follow-up after post-assessment.
  It consist of 5 items that evaluate the frequency and the intensity of anxious symptoms and their interference with the person's work or school life and social life. It is responded on a 5-point Likert scale (0=No anxiety- 4=The worst anxiety possible). The total score range from 0 to 20 points. Higher scores are indicative of greater severity and functional impairment as a result of anxious symptoms. In the Spanish population the clinical cut-off has been stablished in 10 points.
Fertility Problem Inventory (FPI) | Pre-intervention; Post-intervention, 11 weeks from pre-assessment; 1 month follow-up after post-assessment; 3 months follow-up after post-assessment; 6 months follow-up after post-assessment.
  It is composed by 46 items that assess infertility-related stress. It is responded by a 7-points Likert scale (0=completely disagree - 6=completely agree). It is possible to obtain a total score of perceived stress and also it is possible to calculate 5 subscale scores (social concerns, sexual concerns, relationship concerns, need for parenthood and, reject to child-free living). Higher scores indicate greater stress.
Fertility Quality of Life Questionnaire (FertiQoL) | Pre-intervention; Post-intervention, 11 weeks from pre-assessment; 1 month follow-up after post-assessment; 3 months follow-up after post-assessment; 6 months follow-up after post-assessment.
  This instrument is composed by 36 items assessing quality of life during fertility treatments. It is responded by a 5-point Likert scale (0=very bad - 4 = very good). Total scores range from 0 to 136 points, higher global scores indicating greater quality of life.
Difficulties in Emotion Regulation Scale (DERS) | Pre-intervention; Post-intervention, 11 weeks from pre-assessment; 1 month follow-up after post-assessment; 3 months follow-up after post-assessment; 6 months follow-up after post-assessment.
  Consists of 36-item of six dimension of emotion regulation (nonacceptance of emotions, difficulties in engaging in goal-directed behaviours, impulse control difficulties, lack of emotional awareness, limited access to emotion regulation strategies and lack of emotional clarity). Items are rated on a scale of 1 ("almost never [0-10%]") to 5 ("almost always [91-100%]"). Higher scores indicate more difficulties in emotion regulation.
The Multidimensional Emotional Disorder Inventory (MEDI) | Pre-intervention; Post-intervention, 11 weeks from pre-assessment; 1 month follow-up after post-assessment; 3 months follow-up after post-assessment; 6 months follow-up after post-assessment.
  This is a self-report measure that includes 49 items assessing the main transdiagnostic dimensions of Emotional Disorders: Neurotic Temperament; Positive Temperament; Depressed Mood; Autonomic Arousal; Somatic Anxiety; Social Anxiety; Intrusive Cognitions, Traumatic Re-experiencing; Avoidance. It is responded by a 9-point Likert scale (0=not characteristic of me - 8=extremely characteristic of me). Result for each dimension allows to obtain a profile to emotional disorders.
Web-page adherence | Post-intervention (11 weeks from pre-intervention assessment).
  The web automatically records the number of modules completed. At the end of the intervention, the number of modules completed will be analyzed in proportion to the number of modules programmed.
Adaptation of the Client Satisfaction Questionnaire (CSQ-8) | Post-intervention (11 weeks from pre-intervention assessment).
  This adaptation is composed of 7 items assessing (a) quality of the intervention and quality of its components, (b) discomfort experienced during treatment, (c) satisfaction with their participation in an online individual format.
Unified Protocol Satisfaction questionaire | Post-intervention (11 weeks from pre-intervention assessment).
  It consists of 7 questions that assess the general usefulness of the Unified Protocol to improve emotion regulation skills and the specific usefulness of each of the Unified Protocol skills.

CONTACTS AND LOCATIONS:
Locations (1):
- Jorge Osma, Teruel, Spain

IPD SHARING:
Plan to Share IPD: No